CLINICAL TRIAL: NCT05101577
Title: Recurrence Rate of Trigeminal Neuralgia in Patients Treated With Percutaneous Stereotactic Continuous Radiofrequency Rhizotomy at 80 Degrees Celsius for 90 Seconds- a Single Center Study.
Brief Title: Recurrence of Trigeminal Neuralgia in Patient's Undergoing Radiofrequency Ablation
Status: Completed | Type: Observational
Sponsor: Shifa Clinical Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Hasan Wasim, Fellow Pain Medicine, Shifa Clinical Research Center
Other Study IDs: ShifaCRC
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Trigeminal Neuralgia, Idiopathic
Keywords: trigeminal neuralgia; stereotactic rhizotomy; radiofrequency ablation; recurrence
MeSH Terms: conditions — Trigeminal Neuralgia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find recurrence rate of the trigeminal neuralgia after patients undergo stereotactic rhizotomy by radiofrequency ablation at 80 degrees Celsius for 90 seconds under fluoroscopic guidance, a protocol that was modified from the originally described parameters for rhizotomy by John Tew, Chad J. Morgan and Andresw Grande et al. The presumption being that the higher temperature of the probe tip would lead to a more long-lasting lesion and lesser recurrence, but at the cost of more frequent sensory and motor deficits.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients fulfilling ICHD criteria:

Recurrent paroxysms of unilateral facial pain in the distribution(s) of one or more divisions of the trigeminal nerve, with no radiation beyond, and fulfilling criteria B and C

A. Pain has all of the following characteristics:

1. lasting from a fraction of a second to 2 minutes
2. severe intensity
3. electric shock-like, shooting, stabbing or sharp in quality B. Precipitated by innocuous stimuli within the affected trigeminal distribution C. Not better accounted for by another ICHD-3 diagnosis.

2. Age: Adults of both sexes 3. MRI brain ruled out organic or structural pathologies

Exclusion Criteria:

* 1. Patient with concomitant co-morbid conditions like brain tumours, vascular pathologies or coagulopathies.

  2. Patients who had previously undergone trigeminal ganglion neurolysis with either alcohol or phenol.

  3. Patients who were lost to follow-up before the completion of 6-month period or had not visited back after the procedure 4. Patients on oral anticoagulants 5. Patients declared high risk or ASA 3 and above for general anaesthesia.

Ages: 27 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients of all genders presenting to Pain Clinic, referred of otherwise, diagnosed to have trigeminal neuralgia without concomitant central nervous pathologies including space occupying lesions, vascular and auto-immune disorders, who were planned for stereotactic rhizotomy under deep sedation and monitored anesthesia care as daycare cases.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of trigeminal neuralgia after stereotactic rhizotomy | Recurrence within 12 months of the intervention
  Recurrence of pain in the same distribution of the trigeminal nerve branch or branches for which the stereotactic rhizotomy was originally performed
Proportion of patients with neurological deficits after stereotactic rhizotomy | 5 years
  locally deviced protocol for stereotactic rhizotomy of the involved trigeminal gangion dictates the use of higher temperature of 80 degree Celsius for 90 seconds, which translates into better pain relief and longer pain free intervals at the cost of higher percentage of sensory and motor deficits

CONTACTS AND LOCATIONS:
Overall Officials: Salman A. Saleem, MBBS;FCPS, Study Director — Shifa Clinical Research Center

REFERENCES:
- [Background] Taha JM, Tew JM Jr, Buncher CR. A prospective 15-year follow up of 154 consecutive patients with trigeminal neuralgia treated by percutaneous stereotactic radiofrequency thermal rhizotomy. J Neurosurg. 1995 Dec;83(6):989-93. doi: 10.3171/jns.1995.83.6.0989. PMID 7490643
- [Background] Rashid A, Pintea B, Kinfe TM, Surber G, Hamm K, Bostrom JP. LINAC stereotactic radiosurgery for trigeminal neuralgia -retrospective two-institutional examination of treatment outcomes. Radiat Oncol. 2018 Aug 22;13(1):153. doi: 10.1186/s13014-018-1102-2. PMID 30134992
- [Background] Kao CH, Lee MH, Yang JT, Tsai YH, Lin MH. Percutaneous Radiofrequency Rhizotomy Is Equally Effective for Trigeminal Neuralgia Patients with or Without Neurovascular Compression. Pain Med. 2022 Apr 8;23(4):807-814. doi: 10.1093/pm/pnab221. PMID 34264315
- [Background] Zhao G, Sun X, Zhang Z, Yang H, Zheng X, Feng B. Clinical efficacy of MVD combined with PSR in the treatment of primary trigeminal neuralgia. Exp Ther Med. 2020 Aug;20(2):1582-1588. doi: 10.3892/etm.2020.8871. Epub 2020 Jun 10. PMID 32742390
- [Background] Elnashar A, Patel SK, Kurbanov A, Zvereva K, Keller JT, Grande AW. Comprehensive anatomy of the foramen ovale critical to percutaneous stereotactic radiofrequency rhizotomy: cadaveric study of dry skulls. J Neurosurg. 2019 Apr 19;132(5):1414-1422. doi: 10.3171/2019.1.JNS18899. Print 2020 May 1. PMID 31003215